CLINICAL TRIAL: NCT03449719
Title: A 2 Arm, Phase II Controlled Randomized Trial Comparing Efficacy and Safety of Abiraterone and Abiraterone Associated With of Ablative Radiation Therapy in Patients With Oligometastatic Castration Resistant Prostate Cancer (ARTO Trial)
Brief Title: Phase II Randomized Trial of Radiation Therapy in Oligometastatic mCRPC Prostate Cancer (ARTO)
Acronym: ARTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lorenzo Livi (Other)
Responsible Party: Sponsor-Investigator, Lorenzo Livi, Prof, Azienda Ospedaliero-Universitaria Careggi
Organization: Azienda Ospedaliero-Universitaria Careggi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTO
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Rate of PSA Response in Oligometastatic,CRPC Undergoing SBRT in Combination With Abiraterone Acetate (AA), Compared to Patients Treated With AA Alone
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: A Phase II study is suitable to investigate the interaction of systemic therapy (ADT and abiraterone) with locoregional therapy (SBRT). The duration of the study equal to 40 months was defined taking into account both the expected time of occurrence of investigated endpoints and feasibility considerations related to patient availability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abiraterone (Active Comparator): The treatment phase consists of systemic treatment with abiraterone acetate 1000 mg daily and prednisone 10 mg daily, plus GnRH agonist or antagonist (control arm).
  Interventions: Drug: Abiraterone Acetate
- Abiraterone associated withAblative Radiation (Experimental): the patients in the experimental arm will receive SBRT to all metastatic lesions, concomitantly with abiraterone acetate.
  SBRT will be delivered in 1 to 5 fractions, and the dose and fractionation schedule will depend on the size and location of the lesion and the surrounding normal tissue constraints in accordance with AAPM Task Group 101 recommendations.
  Considering an Alfa/beta of 3, a BED3 > 100 Gy is recommended
  Interventions: Radiation: SBRT - Ablative radiation Therapy; Drug: Abiraterone Acetate

INTERVENTIONS:
Radiation: SBRT - Ablative radiation Therapy — The current phase II randomized trial,"Ablative Radiation Therapy in patients with Oligometastatic castration resistant prostate cancer (ARTO trial)" aims to evaluate the difference in PSA response rate between the experimental arm (AA+SBRT) and control arm (AA) in metastatic castration-resistant prostate cancer patients.
  Other Names: AA+SBRT
  Arms: Abiraterone associated withAblative Radiation
Drug: Abiraterone Acetate — systemic treatment with abiraterone acetate 1000 mg daily and prednisone 10 mg daily, plus GnRH agonist or antagonist
  Other Names: AA

SUMMARY:
Metastatic castration resistant prostate cancer causes approximately 258400 deaths annually worldwide.

In the presence of metastatic disease, systemic treatment remains the main clinical option. However, since the introduction of highly sensitive imaging techniques, a new clinical entity of metastatic patients with a limited number of lesions has been defined: oligometastatic patients.

Although a clear benefit has yet to be demonstrated in this group of patients, the use of stereotactic body radiotherapy (SBRT) or other local therapies directed against all active lesions has been suggested as a possible salvage treatment.

Irradiation of metastatic foci may delay the emergence of castration resistance because irradiation is effective against both ADT¬ sensitive and ADT ¬resistant prostate cancer cells as shown in re-biopsy studies. Stereotactic body radiation therapy has been used in this setting to defer the initiation of ADT in patients with oligometastatic prostate cancer with notable results.

Abiraterone acetate is a first class inhibitor of cytochrome P ¬450c17, a critical enzyme in extragonadal and testicular androgen synthesis. Abiraterone plus low dose prednisone improves survival in patients with metastatic castration ¬resistant prostate cancer who have already received docetaxel and the combination therapy has received regulatory approval for this indication. Furthermore, Abiraterone acetate is approved also in patients who did not undergo to docetaxel chemotherapy, after the results from the COU-AA 302 study; Results from this phase III trial confirmed the benefit in chemo-naïve patients treated with abiraterone acetate both in terms of overall and radiological progression free survival, if compared to placebo.

In oligometastatic CRPC, the rationale to use SBRT is that the addition of a local ablative treatment could improve disease control in mCRPC patients treated with a systemic therapy.

The current phase II randomized trial,"Ablative Radiation Therapy in patients with Oligometastatic castration resistant prostate cancer (ARTO trial)" aims to evaluate the difference in PSA response rate between the experimental arm (AA+SBRT) and control arm (AA) in metastatic castration-resistant prostate cancer patients

DETAILED DESCRIPTION:
This phase II randomized trial was designed to evaluate the difference in PSA response rate between the experimental arm (AA+SBRT) and control arm (AA). PSA response will be defined as a post-treatment decrease > 50% from baseline measured within 6 months.

Study design

This is a phase II randomized multicenter study in patients affected by oligo ¬mCRPC, treated with standard of care (GnRH agonist or antagonist plus abiraterone acetate and prednisone) and randomized to receive SBRT to all sites of disease. Patients will be randomly assigned in a 1:1 ratio to both treatment, stratified by Centre, Performance Status, and number of metastases.

Randomization will be performed the same day of the baseline evaluation (+/-3 days).

Planned size of the overall study population is 174 patients, 87 for each arm. The study will include a screening phase and a treatment phase.

The screening phase allows for assessment of subject eligibility, demographics, PSA, testosterone, comorbidities and current drug therapies up to 45 days prior to randomization.

The treatment phase consists of systemic treatment with abiraterone acetate 1000 mg daily and prednisone 10 mg daily, plus GnRH agonist or antagonist (control arm). Furthermore, the patients in the experimental arm will receive SBRT to all metastatic lesions.

SBRT will be delivered in 1 to 5 fractions, and the dose and fractionation schedule will depend on the size and location of the lesion and the surrounding normal tissue constraints in accordance with AAPM Task Group 101 recommendations [19]. Considering an Alfa/beta of 3, a BED3 > 100 Gy is recommended. The total planned duration of the study is 40 months, consisting in 28 months enrollment period, during which patients will perform the screening and will begin standard of care treatment with or without SBRT and later phase of 12 months in which patients will continue the treatment with standard of care and will be submitted to periodic checks every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Each potential subject must satisfy all of the following criteria to be enrolled in the study.

  1. Metastatic disease and only <3 metastatic sites recorded (irrespective if nodal or bone).
  2. Patients should have received abiraterone acetate for 30 days before eventual start of radiotherapy in the experimental arm (+/- 3 days)
  3. Asymptomatic or mildly symptomatic patients according to clinical judgement.
  4. Age ≥ 18 years.
  5. Subject must have signed an informed consent document indicating that they understand the purpose of procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* 1. More than 3 metastatic lesions.

  2. Visceral involvement.

  3. Known or suspected contraindications or hypersensitivity to Abiraterone, GnRH agonist/antagonist or Radiotherapy.

  4. Comorbidities that contraindicate Abiraterone, GnRH agonist/antagonist or Radiotherapy.

  5. Any condition for which, in the option of the investigator, participation would not be in the best interest of subject.

  6. Patients who received previous therapies for mCRPC (excluded hormonal therapy)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male with metastatic castration resistant prostate cancer
Enrollment: 174 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
rate PSA | within 6 months
  rate of PSA response in nodal and/or bone oligometastatic (⩽3 lesions), castration resistant prostate cancer patients undergoing SBRT in combination with AA (experimental arm), compared to patients treated with AA (control arm). PSA response will be defined as a post-treatment decrease > 50% from baseline measured within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, Prof, Principal Investigator — Radioterapia Oncologica AOUC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Francolini G, Allegra AG, Detti B, Di Cataldo V, Caini S, Bruni A, Ingrosso G, D'Angelillo RM, Alitto AR, Augugliaro M, Triggiani L, Parisi S, Facchini G, Banini M, Simontacchi G, Desideri I, Meattini I, Valicenti RK, Livi L; ARTO Working Group members. Stereotactic Body Radiation Therapy and Abiraterone Acetate for Patients Affected by Oligometastatic Castrate-Resistant Prostate Cancer: A Randomized Phase II Trial (ARTO). J Clin Oncol. 2023 Dec 20;41(36):5561-5568. doi: 10.1200/JCO.23.00985. Epub 2023 Sep 21. PMID 37733977
- [Derived] Francolini G, Di Cataldo V, Detti B, Simontacchi G, Loi M, Valzano M, Desideri I, Meattini I, Mangoni M, Livi L. Killing two birds with a stone: how to maximise benefit from metastasis-directed therapy and modern systemic treatment in oligometastatic hormone sensitive prostate cancer. Clin Exp Metastasis. 2022 Dec;39(6):841-843. doi: 10.1007/s10585-022-10187-2. Epub 2022 Oct 15. PMID 36242700
- [Derived] Francolini G, Loi M, Detti B, Desideri I, Mangoni M, Simontacchi G, Meattini I, Livi L. Integrating stereotactic body radiation therapy (SBRT) and systemic treatments in oligoprogressive prostate cancer: new evidence from the literature. Clin Exp Metastasis. 2021 Apr;38(2):227-230. doi: 10.1007/s10585-021-10072-4. Epub 2021 Jan 20. PMID 33471291

DOCUMENTS (1):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03449719/Prot_000.pdf